CLINICAL TRIAL: NCT04955002
Title: Food Choice, Psychological Bias, and Genetic Predisposition
Status: Completed | Type: Observational
Sponsor: Oxford Brookes University (Other)
Collaborators: St. Mary's University, Twickenham (Other)
Responsible Party: Principal Investigator, Catherine Graham, Principle Investigator, Lecturer in Nutrition, Oxford Brookes University
Other Study IDs: 0521_01
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Food Preferences; Genetic Predisposition; Psychological
MeSH Terms: conditions — Food Preferences; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy UK adults: Healthy UK adults
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This project aims to assess if food choice is impacted by loss aversion (LA), and if this differs based on genetic predisposition to LA, in a UK healthy cohort.

DETAILED DESCRIPTION:
Food choice, defined as how individuals decide on what to buy and eat, involves the acceptance and rejection of specific foods. Food customisation is becoming more common amongst food retailers, allowing customers to alter their meals to their preferences by removing or adding items. Today, food choice is viewed as more complex, food choices are not just dictated by taste but nutritional quality, allergens, and habits. For example, the framework provided for food customisation (e.g. pizza with toppings or a build you own pizza) and the perceived 'healthiness' of food items (e.g. the pizza toppings) can alter food choice. Psychological reasoning, the process by which humans make decisions by drawing conclusions can play a role in food choice; however, humans can possess a psychological bias leading to illogical decision making. Genetics can too play a role in decision making resulting in predetermined influence on food choice. This research wishes to determine if individual's genetics can affect their food choices by researching psychological biases to food choices.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no known health condition)
* 18 + years of age
* UK based

Exclusion Criteria:

* Vegetarian
* Vegan
* Other dietary pattern that restricts the consumption of animal products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female, adult (18+), UK-based
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Frequency of food items remaining | December 2021
  Number of food items added/removed from each decision frame
Frequency of healthy and unhealthy items remaining | December 2021
  Number of healthy and unhealthy food items added/removed from each decision frame
Loss aversion score | December 2021
Genotype: BDNF Val/Met (rs6265), and DRD2 ANNKK1 Taq1a/ANKK1 (rs1800497) | December 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Brookes University, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No